CLINICAL TRIAL: NCT02148614
Title: Intake of a Polysaccharides Mix (LibraMedR) in Obese Children. 1. Postprandial Effects on Metabolism, Hormones and Satiety; 2. Effects on Body Fat, Glucide and Fat Metabolism After a 60-day Treatment.
Brief Title: Effects of Intake of a Polysaccharides Mix on Metabolism, Hormones and Satiety in Obese Children.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Claudio Maffeis, MD, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 392CEP
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be randomly assigned to treatment with placebo or LibramedR with a double blind clinical trial.
  Interventions: Drug: Placebo
- Libramed (Active Comparator): Subjects will be randomly assigned to treatment with placebo or LibramedR with a double blind clinical trial.
  Interventions: Drug: Libramed

INTERVENTIONS:
Drug: Placebo — Phase 1. Two tablets in a single preprandial dose Phase 2. Two tablets daily for 60 days
  Other Names: No drug
  Arms: Placebo
Drug: Libramed — Phase 1. Two tablets in a single postprandial dose Phase 2. Two tablets daily for 60 days
  Other Names: Policaptil Gel Retard
  Arms: Libramed

SUMMARY:
AIMS

Phase 1. Verify whether the intake of LibramedR is able to induce a better endocrine and metabolic profile.

Phase 2. Verify whether treatment with LibramedR for 60 days produces a better glycaemic profile after oral glucose load.

SUBJECTS

Will be recruited 80 obese children for phase 1 and 40 obese children for phase 2.

Subjects will be randomly assigned to treatment with placebo or LibramedR with a double blind clinical trial.

METHODS

Experimental protocol phase 1

Each child will arrive at the UOC at 8 a.m., in fasting. A blood sample will be taken. Then patients will be given two LibramedR tablets or placebo. After 20 minutes they will be given a mixed meal (equal to 15 kcal per kg of lean body mass). Blood samples will then be taken at 30-minute intervals for the first two hours and 60 minutes for the following two hours, for the determination of metabolites and hormones for a total of 4 hours. The level of satiety will be quantified through a visual analog scale.

Experimental protocol phase 2

Based on the results of the OGTT performed in recruitment phase, children will be divided into two groups: group A, children with blood glucose 2 hours after oral load higher than the median and group B, children with blood glucose 2 hours after oral load below the median.

The children of group A will be randomly assigned to LibramedR treatment or placebo for 60 days, after which they will repeat Anthropometric measurements, bioelectrical impedance, OGTT and blood chemistry. They will also repeat dietary and sport anamnesis .

During the 60 days, the children of both groups will receive the same dietary treatment consisting of a low-calorie and balanced diet, and recommendations to practice more sport.

Every 15 days a research assistant will contact the families to reinforce treatment adherence.

EXPECTED RESULTS

Phase 1 LibramedR intake should cause a lower increase in postprandial blood glucose, insulin, triglycerides and a greater decrease in ghrelin levels compared to placebo treatment;

Phase 2 The treatment with LibramedR should be associated with a decrease in blood glucose and insulin secretion after OGTT compared to placebo treatment.

DETAILED DESCRIPTION:
INTRODUCTION

The postprandial phase has a fundamental role in metabolic regulation. In fact, being exposed to high levels of substrates such as glucose and fatty acids after food intake tends to increase the risk of cardiovascular disease. This is even more relevant in reference to the amount of hours in which the subject is in postprandial condition and therefore exposed to high concentrated substrates. Food intake, moreover, regulates gastrointestinal secretion of hormones which help balance between hunger and satiety, by regulating nutrients supply and peripheral substrate consumption.

An obese subject, due to excessive body fat and of its accumulation, presents high insulin, glucose and triglyceride blood levels, and blood pressure which increase the risk of cardiovascular disease. Since the body is for most of the time in postprandial phase, substrate and hormone containment a few hours after food intake helps limit exposition to cardiovascular risks and potential metabolic and vascular damage.

On equal food and energy intake, a meal's composition has great influence over postprandial and hormonal metabolic profiles. A high lipid/carbohydrate ratio meal, for instance, produces higher postprandial triglycerides and GLP-1 secretion, and lower glucose and insulin levels than an isocaloric, isoproteic meal with low lipid/carbohydrate ratio. The intake of polysaccharides macromolecules produces an endoluminal gel that reduces and delays the absorption of intestinal nutrients, especially glucose and lipids. The intake of soluble fibre is associated to a better glycaemic profile and postprandial lipemia.

At present, it is not known whether the intake of macromolecules such as Policaptil Gel RetardR polysaccharides (LibramedR) before the meal affects the metabolic response (substrate oxidation, hormonal and circulating nutrients variation) and the satiating effect compared to the same meal after taking placebo, and could therefore help to reduce postprandial cardiovascular risks.

AIMS

Phase 1. Verify whether the intake of LibramedR is able to induce a better endocrine (lower blood insulin and ghrelin postprandial levels) and metabolic (decreasing postprandial glycaemia, fatty acids and triglycerides) profile.

Phase 2. Verify whether treatment with LibramedR for 60 days produces a better glycaemic profile after oral glucose load.

SUBJECTS

The standard clinical practice at the UOC of Diabetology, Clinical Nutrition and Obesity in Children Pediatrics, ULSS 20 Verona for obese children, consists in the medical examination with assessment of the stage of pubertal development, anthropometric measurements (height, weight, waist circumference), bioimpedance analysis of body composition (TanitaR), dietary anamnesis (food diary) and sport anamnesis (hours per day of video exposure and hours per week of sport). On the next day, the patient performs an oral glucose load curve (OGTT), a blood chemistry sampling for the determination of the lipid profile and ALT. These practices, which are common clinical procedures, are not part the present project.

Within this group of patients with these clinical and biochemical characteristics, will be recruited for this study 80 children for phase 1 and 40 children for phase 2.

Phase 1 Inclusion criteria: age (10 + 2 years), ethnicity (Caucasians), obesity (BMI> cut-off of BMI for age and gender indicative of obesity, defined by the International Obesity Task Force), acceptance to take part in the study.

Exclusion criteria: birth defects, genetic disorders, chronic diseases, obesity secondary to chronic intake of drugs or endocrine causes or genetic therapy for obesity already in progress.

Phase 2 Inclusion criteria: age (10 + 2 years), ethnicity (Caucasians), obesity, acceptance to take part in the study, blood glucose levels 2 hours after oral glucose tolerance test (performed prior to recruitment) above the median of reference.

Exclusion criteria: birth defects, genetic disorders, chronic diseases, obesity secondary to chronic intake of drugs or endocrine causes or genetic therapy for obesity already in progress, blood glucose 2 hours after an oral glucose load below the median of reference.

Subjects will be randomly assigned to treatment with placebo or LibramedR with a double blind clinical trial.

METHODS

Experimental protocol phase 1 Each child will arrive at the UOC at 8 a.m., in fasting since 9 p.m. the previous evening. A blood sample will be taken with a needle cannula on the antecubital vein. Then patients will be given two LibramedR tablets or placebo. After another 20 minutes they will be given a mixed meal to be consumed within 20 minutes. Blood samples will then be taken at 30-minute intervals for the first two hours and 60 minutes for the following two hours, for the determination of metabolites and hormones for a total of 4 hours (baseline + 6 blood samples).

Sample meal The child will have a mixed meal equal to 15 kcal per kg of lean body mass, in order to standardize the intake according to their metabolically active mass.

Meal composition: bread, cooked ham, ice cream (stracciatella), water, cheese (PhiladelphiaR).

% of total energy: protein 12.2% carbohydrate 52.6%, lipid 35,2%, fiber 8% (caloric density will be equal to 1.4 kcal/g).

Subjective appetite The level of satiety will be quantified through a visual analog scale simplified for use with children at 30-minute intervals for the first two hours and 60 minutes for the following two hours.

Experimental protocol phase 2 Based on the results of the OGTT performed in recruitment phase, children will be divided into two groups: group A, children with blood glucose 2 hours after oral load higher than the median (lower glucose tolerance) and group B, children with blood glucose 2 hours after oral load below the median (greater glucose tolerance).

The children with a lower glucose tolerance will be randomly assigned to LibramedR treatment or placebo for 60 days (two tablets daily), after which they will repeat Anthropometric measurements, bioelectrical impedance, OGTT and blood chemistry (lipid profile, ALT and HbA1c). They will also repeat dietary and sport anamnesis .

During the 60 days, the children of both groups will receive the same dietary treatment consisting of a low-calorie (less than 30% of the energy requirements estimated by sex, age and height) and balanced (protein = 15%, carbohydrates = 55%, lipids = 30%) diet, and recommendations to change their sedentary lifestyle and practice more sport.

Every 15 days a research assistant will contact the families to reinforce treatment adherence.

STATISTICAL ANALYSIS

Calculating sample size phase 1 The sample size was calculated to detect a difference of at least 300 mg / dl * 240 min. AUC glucose measured between the zero and 240 minutes after taking the test between the groups that received LibramedR before the meal and the one that took placebo, with 85% power and 5% alpha error. The mean and standard deviation of the glucose AUC group who received placebo were obtained from a previous study carried out by our group (C Maffeis et al. vs. A High-Fat. in Moderate-fat Meal in Obese Boys: Nutrient Balance, Appetite, and Gastrointestinal Hormone Changes, Obesity 2010; 18 (3) :449-55). The average value of the group taking LibramedR was 8% lower than the placebo group, while the standard deviation was supposedly equal to that of the group who took placebo.

Calculating sample size phase 2 The sample size was calculated to detect a difference of 2100 mg / dl * min. of glucose AUC measured between 0 and 120 minutes after an oral glucose load in the group treated with LibramedR and the placebo group, with 90% power and 5% alpha error. The mean and standard deviation of the AUC glucose placebo arm were taken from our internal database of 100 patients who performed a glucose tolerance curve and the arm's standard deviation with LibramedR was supposedly equal to that of the other arm.

Statistical analysis phase 1 The mean values of the physical, biochemical and metabolic variables and area under the curve (AUC) of metabolites and hormones of children who have taken LibramedR will be compared with Student's t test for two-tailed unpaired data with those children who have taken the placebo, or with non-parametric test, if specified. Postprandial metabolic and hormonal parameter changes in the two groups will be compared with ANOVA repeated measures.

The SPSS 21.0 software will be used to perform the analysis. The level of significance of the test will be set at p <0.05.

Statistical analysis phase 2 In each group, average physical, biochemical and metabolic variables and area under the curve (AUC) glucose and insulin values at recruitment (baseline) will be compared with follow-up values, with Student's t tests for paired data, or non-parametric tests, if specified. The comparison between the delta of the variables measured at baseline and follow-up for the group treated with LibramedR and the placebo group will be performed with Student's t test with two queues for unpaired data or with non-parametric test, if specified. Hormonal and metabolic parameters change during afterload of glucose in the two groups will be compared with ANOVA for repeated measures.

The software SPSS 21.0 will be used to perform the analysis. The level of significance of the test will be set at p <0.05.

EXPECTED RESULTS

Protocol phase 1 LibramedR intake should cause a lower increase in postprandial blood glucose, insulin, triglycerides and a greater decrease in ghrelin levels compared to placebo treatment;

Protocol phase 2 The treatment with LibramedR should be associated with a decrease in blood glucose and insulin secretion after OGTT compared to placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* age, ethnicity (Caucasians), obesity (BMI> cut-off of BMI for age and gender indicative of obesity, defined by the International Obesity Task Force), acceptance to take part in the study.

Exclusion criteria:

* birth defects, genetic disorders, chronic diseases, obesity secondary to chronic intake of drugs or endocrine causes or genetic therapy for obesity already in progress.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2014-01; Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve of plasma glucose. | Meal test 4-hours frame time
  Both placebo and intervention subjects will undergo a 4 hours lasting meal test during which blood glucose will be measured periodically and the area under the curve of plasma glucose during the test period will be then calculated for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Maffeis, MD, Principal Investigator — Pediatric Diabetes and Metabolic Disorders Unit, Department of Life and Reproduction Sciences, University of Verona
Locations (1):
- Pediatric Diabetes and Metabolic Disorders Unit, Department of Life and Reproduction Sciences, University of Verona, 1 Piazzale Stefani, Verona, Italy

REFERENCES:
- [Background] Alipour A, Elte JW, van Zaanen HC, Rietveld AP, Castro Cabezas M. Novel aspects of postprandial lipemia in relation to atherosclerosis. Atheroscler Suppl. 2008 Sep;9(2):39-44. doi: 10.1016/j.atherosclerosissup.2008.05.007. Epub 2008 Jul 1. PMID 18595782
- [Background] Murphy KG, Bloom SR. Gut hormones and the regulation of energy homeostasis. Nature. 2006 Dec 14;444(7121):854-9. doi: 10.1038/nature05484. PMID 17167473
- [Background] Shay CM, Ning H, Daniels SR, Rooks CR, Gidding SS, Lloyd-Jones DM. Status of cardiovascular health in US adolescents: prevalence estimates from the National Health and Nutrition Examination Surveys (NHANES) 2005-2010. Circulation. 2013 Apr 2;127(13):1369-76. doi: 10.1161/CIRCULATIONAHA.113.001559. Epub 2013 Apr 1. PMID 23547177
- [Background] Maffeis C, Surano MG, Cordioli S, Gasperotti S, Corradi M, Pinelli L. A high-fat vs. a moderate-fat meal in obese boys: nutrient balance, appetite, and gastrointestinal hormone changes. Obesity (Silver Spring). 2010 Mar;18(3):449-55. doi: 10.1038/oby.2009.271. Epub 2009 Aug 27. PMID 19713952
- [Background] Verbeke K, Ferchaud-Roucher V, Preston T, Small AC, Henckaerts L, Krempf M, Wang H, Vonk RJ, Priebe MG. Influence of the type of indigestible carbohydrate on plasma and urine short-chain fatty acid profiles in healthy human volunteers. Eur J Clin Nutr. 2010 Jul;64(7):678-84. doi: 10.1038/ejcn.2010.92. Epub 2010 May 26. PMID 20502475